CLINICAL TRIAL: NCT01529541
Title: A Multicenter, Randomized, Double-blind, Double Dummy, Active-controlled, Therapeutic Confirmatory Trial(Phase 3) to Evaluate the Efficacy and Safety of CWP-0403 Compared With Sitagliptin Added to Ongoing Metformin Therapy in Patients With Type 2 DM Insufficiently Controlled With Metformin Alone
Brief Title: Efficacy and Safety of CWP-0403 Compared to Sitagliptin in Patients With Type 2 Diabetes Mellitus Insufficiently Controlled With Metformin Alone
Acronym: CWP-DIANA-302
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CWP-DIANA-302
Record Dates: First submitted 2012-02-06; First posted 2012-02-09 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: CWP-0403; Sitagliptin; Metformin; type 2 DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — anagliptin; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin (Active Comparator): Sitagliptin 100mg
  Interventions: Drug: Sitagliptin
- CWP-0403 (Experimental): CWP-0403 100mg
  Interventions: Drug: Anagliptin

INTERVENTIONS:
Drug: Anagliptin — Anagliptin 100mg, tablet, twice a day (BID)
  Arms: CWP-0403
Drug: Sitagliptin — Sitagliptin 100mg, tablet, once a day (QD)
  Arms: Sitagliptin

SUMMARY:
This trial is to evaluate the efficacy and safety of CWP-0403 compared to Sitagliptin by proving non-inferiority in patients with type 2 Diabetes Mellitus insufficiently controlled with metformin alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had diagnosed with type 2 DM before 3 months
* Men and women between the age of ≥ 19 and ≤ 75 years
* FPG ≤ 270 mg/dL at screening visit
* Patients who consent to participate in this trial by written Informed Consent Form

Exclusion Criteria:

* Type 1 DM or secondary diabetes
* Subjects who are administrating oral anti-hyperglycemic drugs or have to take a medicine
* Body mass index < 20 kg/m2 or > 40.0kg/m2
* Subjects who are assessed to be inappropriate for this trial by investigator

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The Change in HbA1c from baseline to week24. | 0wk, 8wk, 16wk, 24wk

SECONDARY OUTCOMES:
The proportion of subjects achieving HbA1c<7% at week24 | 0wk, 8wk, 16wk, 24wk
The proportion of subjects achieving HbA1c<6.5% at week24 | 0wk, 8wk, 16wk, 24wk
The change from baseline to week 24: Fasting plasma glucose | 0wk, 24wk
change from baseline to week 24: Fasting serum insulin | 0wk, 24 wk
change from baseline to week 24 in Fasting serum pro-insulin | 0wk, 24wk
change from baseline to week 24 in Fasting serum c-peptide | 0wk, 24wk
change from baseline to week 24 in HOMA-β | 0wk, 24 wk
change from baseline to week 24 in HOMA-IR | 0wk, 24 wk

CONTACTS AND LOCATIONS:
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea